CLINICAL TRIAL: NCT00416065
Title: PET/CT to Identify "Vulnerable" Arterial Plaque
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: plaqueCTIL
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Device: PET/CT imaging

SUMMARY:
The purpose of this research is to evaluate the presence, location and intensity of FDG uptake in the large arteries using the new technology of fused PET/CT imaging and to compare FDG uptake with the presence of arterial calcifications as seen on the simultaneously acquired CT, in order to determine if FDG was increases incalcified plaque or in a different location in the arterial wall. we will also evaluate the relationship between FDG localization and future cardiovascular events in out patient population

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for clinical FDG-PET/CT studies
* Patients 50 yr or older
* Patients signed informed consent

Exclusion Criteria:

* Patients unable or unwilling to tolerate the scan until its completion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2004-04

PRIMARY OUTCOMES:
the impact of the imaging modality on patient management

SECONDARY OUTCOMES:
the impact of the imaging modality on patient management

CONTACTS AND LOCATIONS:
Overall Officials: Ora Israel, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel